CLINICAL TRIAL: NCT05568212
Title: Phase II, Two-cohorts, Randomized Trial Comparing Standard of Care Versus Immune- Based Combination in Relapsed Stage III Non-small-cell Lung Cancer (NSCLC) Pretreated With Chemoradiotherapy and Durvalumab (MEDI4736)
Brief Title: Randomized Trial Comparing Standard of Care Versus Immune- Based Combination in Relapsed Stage III Non-small-cell Lung Cancer (NSCLC) Pretreated With Chemoradiotherapy and Durvalumab
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fondazione Ricerca Traslazionale (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CONDOR
Record Dates: First submitted 2022-06-08; First posted 2022-10-05 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Non-small-cell Lung Cancer Patients
MeSH Terms: interventions — durvalumab; olaparib

STUDY DESIGN:
Intervention Model Description: In the group of individuals progressing during durvalumab theray, patients will be randomized to the experimental arm (durvalumab+chemotherapy) or to the standard arm (chemotherapy alone). The standard arm will act as a calibration arm.
  In the second groups patients will be randomized to the experimental arm durvalumab+chemotherapy followed by maintenance durvalumab+olaparib or to the other experimental arm durvalumab+chemotherapy followed by maintenance durvalumab.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- ARM A (experimental arm) (Experimental): Investigator's choice single-agent chemotherapy plus durvalumab 1500 mg every 3 weeks.
  Interventions: Drug: Durvalumab; Drug: Single-agent chemotherapy
- ARM B (standard arm) (Experimental): Investigator's choice single-agent chemotherapy.
  Interventions: Drug: Single-agent chemotherapy
- ARM C (Experimental): Investigator's choice platinum doublet chemotherapy plus durvalumab 1500 mg every 3 weeks for 4 cycles followed by maintenance durvalumab 1500 mg every 3 weeks plus olaparib 300 mg twice daily.pp
  Interventions: Drug: Durvalumab; Drug: Olaparib tablet; Drug: Platinum doublet chemotherapy
- ARM D (experimental arm) (Experimental): Investigator's choice platinum doublet chemotherapy plus durvalumab 1500 mg every 3 weeks for 4 cycles followed by maintenance durvalumab 1500 mg every 3 weeks
  Interventions: Drug: Durvalumab; Drug: Platinum doublet chemotherapy

INTERVENTIONS:
Drug: Durvalumab — Durvalumab concentrate for solution for infusion will be supplied in glass vials containing 500 mg durvalumab at a concentration of 50 mg/mL
  Arms: ARM A (experimental arm); ARM C; ARM D (experimental arm)
Drug: Olaparib tablet — Olaparib tablets (100 mg and 150 mg strengths) supplied in high-density polyethylene (HDPE) bottles.
  Arms: ARM C
Drug: Single-agent chemotherapy — Investigator's choice single-agent chemotherapy regimen
  Arms: ARM A (experimental arm); ARM B (standard arm)
Drug: Platinum doublet chemotherapy — Investigator's choice platinum doublet chemotherapy
  Arms: ARM C; ARM D (experimental arm)

SUMMARY:
This is a randomized, non-comparative, phase II study investigating whether: 1) the addition of durvalumab to investigator's choice second line chemotherapy prolongs survival versus investigator's choice second line chemotherapy in NSCLC patients with locally advanced disease progressing on durvalumab given after concomitant chemoradiotherapy; 2) whether the addition of olaparib to durvalumab improves survival over durvalumab alone after induction chemoimmunotherapy in patients relapsing after completing durvalumab maintenance therapy for stage III disease.

After evaluation of inclusion and exclusion criteria and after consent form signature, all eligible patients progressing during durvalumab therapy will be in the Part A of the trial randomized to in a 1:1 ratio to investigator's choice single-agent chemotherapy plus durvalumab (Arm A: experimental arm) or to investigator's choice single-agent chemotherapy (Arm B: standard arm). In the clinical trial's Part B, patients progressing after completion of durvalumab therapy will be further randomized in a 1:1.7 ratio to investigator's choice platinum doublet chemotherapy plus durvalumab for 4 cycles followed by maintenance durvalumab plus olaparib (Arm C: experimental arm) or to investigator's choice platinum doublet chemotherapy plus durvalumab for 4 cycles followed by durvalumab (Arm D: experimental arm). Therapy will be continued up to disease progression, toxicity or patient refusal.

ELIGIBILITY:
Inclusion Criteria:

1. Body weight >30kg
2. Recurrent or metastatic NSCLC relapsed during or after completion of chemoradiotherapy with curative intent and maintenance durvalumab for stage III disease. Patients are eligible if they receive at least two cycles of platinum based chemotherapy or radical radiotherapy
3. Tumor tissue available for biomarker testing.
4. Evidence of disease progression during durvalumab maintenance or at the end of planned treatment. Patients who have interrupted planned durvalumab treatment after at least 6 months for reasons other than toxicity or progression (e.g. patient's choice, logistic reasons, intercurrent acute illnesses) are eligible. Patients progressing during the first three months of Durvalumab are not eligible
5. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
6. Patient is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up
7. Age >18 years at time of study entry
8. Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol. Written informed consent and any locally required authorization obtained from the patient/legal representative prior to performing any protocol-related procedures, including screening evaluations.
9. Life expectancy of at least 16 weeks
10. Patients must have normal organ and bone marrow function measured within 28 days prior to administration of study treatment as defined below::

    * Haemoglobin ≥10.0 g/dL with no blood transfusion in the past 28 days
    * Absolute neutrophil count (ANC) ≥1.5 × 109 /L
    * Platelet count ≥100 × 109/L
    * Serum bilirubin ≤1.5 x institutional upper limit of normal (ULN). This will not apply to patients with confirmed Gilbert's syndrome (persistent or recurrent hyperbilirubinemia that is predominantly unconjugated in the absence of hemolysis or hepatic pathology), who will be allowed only in consultation with their physician.
    * AST (SGOT)/ALT (SGPT) ≤2.5 x institutional upper limit of normal unless liver metastases are present, in which case it must be ≤5x ULN
    * creatinine clearance estimated of ≥51 mL/min using the Cockcroft-Gault equation or based on a 24 hour urine test:

    Males:

    Creatinine CL = Weight (kg) x (140 - Age) (mL/min) ---------------------------------------- 72 x serum creatinine (mg/dL)

    Females:

    Creatinine CL = Weight (kg) x (140 - Age) (mL/min) ----------------------------------------- x 0.85 72 x serum creatinine (mg/dL)
11. Female patients should be using adequate contraceptive measures (highly effective method of contraception are present in table 3 of protocol "Highly Effective Methods of Contraception (<1% Failure Rate)"), should not be breastfeeding, from the time of screening throughout the total duration of the drug treatment and the drug washout period (90 days after the last dose of durvalumab monotherapy) or for at least 1 month after last dose of olaparib, or they must totally/truly abstain from any form of sexual intercourse. Females of childbearing potential are defined as those who are not surgically sterile (ie, bilateral salpingectomy, bilateral oophorectomy, or complete hysterectomy) or post-menopausal.
12. Postmenopausal or evidence of non-childbearing status for women of childbearing potential: negative urine or serum pregnancy test within 28 days of study treatment and confirmed prior to treatment on day 1.

    Postmenopausal is defined as:
    * Amenorrheic for 1 year or more following cessation of exogenous hormonal treatments
    * Luteinizing hormone (LH) and Follicle stimulating hormone (FSH) levels in the post menopausal range for women under 50
    * radiation-induced oophorectomy with last menses >1 year ago
    * chemotherapy-induced menopause with >1 year interval since last menses
    * surgical sterilisation (bilateral oophorectomy or hysterectomy)

    The following age-specific requirements apply:
    * Women <50 years of age would be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of exogenous hormonal treatments and if they have luteinizing hormone and follicle-stimulating hormone levels in the post-menopausal range for the institution.
    * Women ≥50 years of age would be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of all exogenous hormonal treatments, had radiation-induced menopause with last menses >1 year ago, had chemotherapy-induced menopause with last menses >1 year ago.
13. Male patients must use a condom during treatment and for 3 months after the last dose of olaparib when having sexual intercourse with a pregnant woman or with a woman of childbearing potential. Female partners of male patients should also use a highly effective form of contraception if they are of childbearing potential. Male patients should not donate sperm throughout the period of taking olaparib and for 3 months following the last dose of Olaparib.

Exclusion Criteria:

1. No evidence of disease progression
2. Patients receiving any systemic chemotherapy or radiotherapy (except for palliative reasons) within 3 weeks prior to study treatment
3. Patients not pretreated with durvalumab with curative intent
4. Patients treated with non-radical radiotherapy or with non conventional radiotherapy
5. More than 4 cycles of platinum-based chemotherapy
6. Rapid progressors. Progressors within first 3 month of treatment will be excluded from this trial
7. Any clinical reason that makes the patient ineligible to receive any investigator's choice single-agent chemotherapy regimen (for patients enrolled in cohorts A and B)
8. Any clinical reason that makes the patient ineligible to receive any investigator's choice platinum-based doublet chemotherapy regimen (for patients enrolled in cohorts C and D)
9. Persistent toxicities (>Common Terminology Criteria for Adverse Event (CTCAE) grade 2) caused by previous cancer therapy, excluding alopecia.
10. Patients with myelodysplastic syndrome/acute myeloid leukaemia or with features suggestive of MDS/AML.
11. Disease progression within the first three months of Durvalumab therapy
12. Tumor tissue not available
13. Evidence of EGFR mutations or ALK or ROS1 rearrangements
14. Performance status >1 (ECOG)
15. Brain metastases are allowed if asymptomatic and pretreated. A scan to confirm the absence of brain metastases is not required. The patient can receive a stable dose of corticosteroids before and during the study as long as these were started at least 4 weeks prior to treatment.
16. Diagnosis of another cancer in the last 3 years, except for in situ carcinoma of cervix, breast and bladder or skin carcinoma (squamous or basaloid)
17. Patient with spinal cord compression unless considered to have received definitive treatment for this and evidence of clinically stable disease for 28 days prior to enrolment..
18. Leptomeningeal disease.
19. Resting ECG indicating uncontrolled, potentially reversible cardiac conditions, as judged by the investigator (eg., unstable ischemia, uncontrolled symptomatic arrhythmia, congestive heart failure, QTcF prolongation >500 ms, electrolyte disturbances, etc.), or patients with congenital long QT syndrome.
20. Uncontrolled pleural effusion, pericardial effusion, or ascites requiring recurrent drainage procedures (once monthly or more frequently). Patients with indwelling catheters (e.g., PleurX) are allowed.
21. Malignancies other than NSCLC within 5 years prior to enrollment, with the exception of those with a negligible risk of metastasis or death (e.g., expected 5-year OS> 90%) treated with expected curative outcome (such as adequately treated carcinoma in situ of the cervix, basal or squamous cell skin cancer, localized prostate cancer treated surgically with curative intent, ductal carcinoma in situ treated surgically with curative intent, grade 1 endometrial carcinoma)
22. History of severe allergic, anaphylactic, or other hypersensitivity reactions to chimeric or humanized antibodies or fusion proteins and patient with a known hypersensitivity to olaparib or any of the excipient of the product.
23. Known hypersensitivity or allergy to any component of the Durvalumab formulation
24. History of autoimmune disease, including but not limited to myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, p psoriatic arthritis, inflammatory bowel disease, vascular thrombosis associated with antiphospholipid syndrome, Wegener granulomatosis, Sjögren's syndrome, Guillain- Barré syndrome, multiple sclerosis, vasculitis, or glomerulonephritis. Patients with: 1) history of autoimmune-related hypothyroidism on a stable dose of thyroid replacement hormone, 2) controlled Type I diabetes mellitus who are receiving a stable dose of insulin regimen and 3) eczema, psoriasis, lichen simplex chronicus of vitiligo with dermatologic manifestations only in less than 10% of body surface area, well controlled at baseline and only requiring low potency topical steroids are eligible for this study.
25. Patients considered a poor medical risk due to a serious, uncontrolled medical disorder, non-malignant systemic disease or active, uncontrolled infection. Examples include, but are not limited to, uncontrolled ventricular arrhythmia, recent (within 3 months) myocardial infarction, uncontrolled major seizure disorder, unstable spinal cord compression, superior vena cava syndrome, extensive interstitial bilateral lung disease on High Resolution Computed Tomography (HRCT) scan or any psychiatric disorder that prohibits obtaining informed consent.
26. Patients unable to swallow orally administered medication and patients with gastrointestinal disorders likely to interfere with absorption of the study medication.
27. History of idiopathic pulmonary fibrosis, organizing pneumonia (e.g., bronchiolitis obliterans), drug-induced pneumonitis, idiopathic pneumonitis, or evidence of active pneumonitis on screening chest CT scan. History of radiation pneumonitis in the radiation field (fibrosis) is permitted.
28. Positive test for HIV
29. Patients with active hepatitis B (chronic or acute; defined as having a positive hepatitis B surface antigen [HBsAg] test at screening) or hepatitis C. Patients with past hepatitis B virus (HBV) infection or resolved HBV infection (defined as the presence of hepatitis B core antibody [HBc Ab] and absence of HBsAg) are eligible. HBV DNA must be obtained in these patients prior to randomization. Patients positive for hepatitis C virus (HCV) antibody are eligible only if PCR is negative for HCV RNA.
30. Active tuberculosis
31. Concomitant use of known strong CYP3A inhibitors (eg. itraconazole, telithromycin, clarithromycin, protease inhibitors boosted with ritonavir or cobicistat, indinavir, saquinavir, nelfinavir, boceprevir, telaprevir) or moderate CYP3A inhibitors (eg.

    ciprofloxacin, erythromycin, diltiazem, fluconazole, verapamil). The required washout period prior to starting study treatment is 2 weeks.
32. Concomitant use of known strong (eg. phenobarbital, enzalutamide, phenytoin, rifampicin, rifabutin, rifapentine, carbamazepine, nevirapine and St John's Wort ) or moderate CYP3A inducers (eg. bosentan, efavirenz, modafinil). The required washout period prior to starting study treatment is 5 weeks for enzalutamide or phenobarbital and 3 weeks for other agents.
33. Major surgery within 2 weeks of starting study treatment and patients must have recovered from any effects of any major surgery.
34. Previous allogenic bone marrow transplant or double umbilical cord blood transplantation (dUCBT).
35. Pregnancy or breast feeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 176 (Estimated)
Dates: Start 2022-05-02 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Overall survival (OS) | 12 months
  Overall Survival (OS) rate at 12 months in patients treated in arm A versus B and in patients treated in arm C versus arm D.

SECONDARY OUTCOMES:
Progression-free survival (PFS) | 12 months
  Progression free survival (PFS) will be calculated from the date of randomization to the first documented evidence of progressive disease or death due to any cause (whichever occurs first) in patients treated in arm A versus B and in patients treated in arm C versus arm D.
Objective response rate (ORR) | Tumor assessment will be performed every 6 weeks for the first 24 weeks and then every 12 weeks until confirmed objective disease progression/death (whichever comes first) assessed up to 30 months.
  Objective response rate (ORR) is defined as the number of subjects with a best overall response (BOR) of CR or PR divided by the number of randomized subjects for each treatment in each coort.
Safety and Incidence of AEs | 39 months
  All adverse events will be reported until 30 days after the final dose of study treatment or until initiation of new systemic anti-cancer therapy, whichever occurs first, and serious adverse events and adverse events of special interest will continue to be reported until 90 days after the final dose of study treatment or until initiation of new systemic anti-cancer therapy, whichever occurs first.
Progression-free survival (PFS) and Overall survival (OS) | 12 months
  Progression-free survival (PFS) and Overall survival (OS) will be evaluated according to biomarkers ((i.e., PD-L1, ERCC1, SLFN11, STK11, KEAP1, p53 expression, DNA repair genes [including BRCA 1-2 mutations] and tumor mutational burden).

CONTACTS AND LOCATIONS:
Overall Officials: Federico Cappuzzo, MD, Principal Investigator — Istituto Nazionale Tumori Regina Elena
Locations (1):
- Istituti Fisioterapici Ospitalieri- Ifo - Istituto Regina Elena, Roma, RM, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Alexandrov LB, Nik-Zainal S, Wedge DC, Aparicio SA, Behjati S, Biankin AV, Bignell GR, Bolli N, Borg A, Borresen-Dale AL, Boyault S, Burkhardt B, Butler AP, Caldas C, Davies HR, Desmedt C, Eils R, Eyfjord JE, Foekens JA, Greaves M, Hosoda F, Hutter B, Ilicic T, Imbeaud S, Imielinski M, Jager N, Jones DT, Jones D, Knappskog S, Kool M, Lakhani SR, Lopez-Otin C, Martin S, Munshi NC, Nakamura H, Northcott PA, Pajic M, Papaemmanuil E, Paradiso A, Pearson JV, Puente XS, Raine K, Ramakrishna M, Richardson AL, Richter J, Rosenstiel P, Schlesner M, Schumacher TN, Span PN, Teague JW, Totoki Y, Tutt AN, Valdes-Mas R, van Buuren MM, van 't Veer L, Vincent-Salomon A, Waddell N, Yates LR; Australian Pancreatic Cancer Genome Initiative; ICGC Breast Cancer Consortium; ICGC MMML-Seq Consortium; ICGC PedBrain; Zucman-Rossi J, Futreal PA, McDermott U, Lichter P, Meyerson M, Grimmond SM, Siebert R, Campo E, Shibata T, Pfister SM, Campbell PJ, Stratton MR. Signatures of mutational processes in human cancer. Nature. 2013 Aug 22;500(7463):415-21. doi: 10.1038/nature12477. Epub 2013 Aug 14. PMID 23945592
- [Background] Apetoh L, Ladoire S, Coukos G, Ghiringhelli F. Combining immunotherapy and anticancer agents: the right path to achieve cancer cure? Ann Oncol. 2015 Sep;26(9):1813-1823. doi: 10.1093/annonc/mdv209. Epub 2015 Apr 28. PMID 25922066
- [Background] Botticella A, Mezquita L, Le Pechoux C, Planchard D. Durvalumab for stage III non-small-cell lung cancer patients: clinical evidence and real-world experience. Ther Adv Respir Dis. 2019 Jan-Dec;13:1753466619885530. doi: 10.1177/1753466619885530. PMID 31686616
- [Background] Brahmer JR, Tykodi SS, Chow LQ, Hwu WJ, Topalian SL, Hwu P, Drake CG, Camacho LH, Kauh J, Odunsi K, Pitot HC, Hamid O, Bhatia S, Martins R, Eaton K, Chen S, Salay TM, Alaparthy S, Grosso JF, Korman AJ, Parker SM, Agrawal S, Goldberg SM, Pardoll DM, Gupta A, Wigginton JM. Safety and activity of anti-PD-L1 antibody in patients with advanced cancer. N Engl J Med. 2012 Jun 28;366(26):2455-65. doi: 10.1056/NEJMoa1200694. Epub 2012 Jun 2. PMID 22658128
- [Background] Butte MJ, Keir ME, Phamduy TB, Sharpe AH, Freeman GJ. Programmed death-1 ligand 1 interacts specifically with the B7-1 costimulatory molecule to inhibit T cell responses. Immunity. 2007 Jul;27(1):111-22. doi: 10.1016/j.immuni.2007.05.016. Epub 2007 Jul 12. PMID 17629517
- [Background] Dunn GP, Old LJ, Schreiber RD. The three Es of cancer immunoediting. Annu Rev Immunol. 2004;22:329-60. doi: 10.1146/annurev.immunol.22.012703.104803. PMID 15032581
- [Background] Ellis S, Carroll KJ, Pemberton K. Analysis of duration of response in oncology trials. Contemp Clin Trials. 2008 Jul;29(4):456-65. doi: 10.1016/j.cct.2007.10.008. Epub 2007 Nov 12. PMID 18187370
- [Background] Escudier B, Motzer RJ, Sharma P, Wagstaff J, Plimack ER, Hammers HJ, Donskov F, Gurney H, Sosman JA, Zalewski PG, Harmenberg U, McDermott DF, Choueiri TK, Richardet M, Tomita Y, Ravaud A, Doan J, Zhao H, Hardy H, George S. Treatment Beyond Progression in Patients with Advanced Renal Cell Carcinoma Treated with Nivolumab in CheckMate 025. Eur Urol. 2017 Sep;72(3):368-376. doi: 10.1016/j.eururo.2017.03.037. Epub 2017 Apr 12. PMID 28410865
- [Background] Gandara DR, von Pawel J, Mazieres J, Sullivan R, Helland A, Han JY, Ponce Aix S, Rittmeyer A, Barlesi F, Kubo T, Park K, Goldschmidt J, Gandhi M, Yun C, Yu W, Matheny C, He P, Sandler A, Ballinger M, Fehrenbacher L. Atezolizumab Treatment Beyond Progression in Advanced NSCLC: Results From the Randomized, Phase III OAK Study. J Thorac Oncol. 2018 Dec;13(12):1906-1918. doi: 10.1016/j.jtho.2018.08.2027. Epub 2018 Sep 11. PMID 30217492
- [Background] Hirano F, Kaneko K, Tamura H, Dong H, Wang S, Ichikawa M, Rietz C, Flies DB, Lau JS, Zhu G, Tamada K, Chen L. Blockade of B7-H1 and PD-1 by monoclonal antibodies potentiates cancer therapeutic immunity. Cancer Res. 2005 Feb 1;65(3):1089-96. PMID 15705911
- [Background] Iwai Y, Ishida M, Tanaka Y, Okazaki T, Honjo T, Minato N. Involvement of PD-L1 on tumor cells in the escape from host immune system and tumor immunotherapy by PD-L1 blockade. Proc Natl Acad Sci U S A. 2002 Sep 17;99(19):12293-7. doi: 10.1073/pnas.192461099. Epub 2002 Sep 6. PMID 12218188
- [Background] Keir ME, Butte MJ, Freeman GJ, Sharpe AH. PD-1 and its ligands in tolerance and immunity. Annu Rev Immunol. 2008;26:677-704. doi: 10.1146/annurev.immunol.26.021607.090331. PMID 18173375
- [Background] Long GV, Weber JS, Larkin J, Atkinson V, Grob JJ, Schadendorf D, Dummer R, Robert C, Marquez-Rodas I, McNeil C, Schmidt H, Briscoe K, Baurain JF, Hodi FS, Wolchok JD. Nivolumab for Patients With Advanced Melanoma Treated Beyond Progression: Analysis of 2 Phase 3 Clinical Trials. JAMA Oncol. 2017 Nov 1;3(11):1511-1519. doi: 10.1001/jamaoncol.2017.1588. PMID 28662232
- [Background] Narwal R, Roskos LK, Robbie GJ. Population pharmacokinetics of sifalimumab, an investigational anti-interferon-alpha monoclonal antibody, in systemic lupus erythematosus. Clin Pharmacokinet. 2013 Nov;52(11):1017-27. doi: 10.1007/s40262-013-0085-2. PMID 23754736
- [Background] Ng CM, Lum BL, Gimenez V, Kelsey S, Allison D. Rationale for fixed dosing of pertuzumab in cancer patients based on population pharmacokinetic analysis. Pharm Res. 2006 Jun;23(6):1275-84. doi: 10.1007/s11095-006-0205-x. Epub 2006 May 26. PMID 16715358
- [Background] Okudaira K, Hokari R, Tsuzuki Y, Okada Y, Komoto S, Watanabe C, Kurihara C, Kawaguchi A, Nagao S, Azuma M, Yagita H, Miura S. Blockade of B7-H1 or B7-DC induces an anti-tumor effect in a mouse pancreatic cancer model. Int J Oncol. 2009 Oct;35(4):741-9. doi: 10.3892/ijo_00000387. PMID 19724910
- [Background] Pardoll DM. The blockade of immune checkpoints in cancer immunotherapy. Nat Rev Cancer. 2012 Mar 22;12(4):252-64. doi: 10.1038/nrc3239. PMID 22437870
- [Background] Paterson AM, Brown KE, Keir ME, Vanguri VK, Riella LV, Chandraker A, Sayegh MH, Blazar BR, Freeman GJ, Sharpe AH. The programmed death-1 ligand 1:B7-1 pathway restrains diabetogenic effector T cells in vivo. J Immunol. 2011 Aug 1;187(3):1097-105. doi: 10.4049/jimmunol.1003496. Epub 2011 Jun 22. PMID 21697456
- [Background] Paz-Ares L, Luft A, Vicente D, Tafreshi A, Gumus M, Mazieres J, Hermes B, Cay Senler F, Csoszi T, Fulop A, Rodriguez-Cid J, Wilson J, Sugawara S, Kato T, Lee KH, Cheng Y, Novello S, Halmos B, Li X, Lubiniecki GM, Piperdi B, Kowalski DM; KEYNOTE-407 Investigators. Pembrolizumab plus Chemotherapy for Squamous Non-Small-Cell Lung Cancer. N Engl J Med. 2018 Nov 22;379(21):2040-2051. doi: 10.1056/NEJMoa1810865. Epub 2018 Sep 25. PMID 30280635
- [Background] Powles T, Eder JP, Fine GD, Braiteh FS, Loriot Y, Cruz C, Bellmunt J, Burris HA, Petrylak DP, Teng SL, Shen X, Boyd Z, Hegde PS, Chen DS, Vogelzang NJ. MPDL3280A (anti-PD-L1) treatment leads to clinical activity in metastatic bladder cancer. Nature. 2014 Nov 27;515(7528):558-62. doi: 10.1038/nature13904. PMID 25428503
- [Background] Qiao M, Jiang T, Ren S, Zhou C. Combination Strategies on the Basis of Immune Checkpoint Inhibitors in Non-Small-Cell Lung Cancer: Where Do We Stand? Clin Lung Cancer. 2018 Jan;19(1):1-11. doi: 10.1016/j.cllc.2017.06.005. Epub 2017 Jun 23. PMID 28716463
- [Background] Ricciuti B, Genova C, Bassanelli M, De Giglio A, Brambilla M, Metro G, Baglivo S, Dal Bello MG, Ceribelli A, Grossi F, Chiari R. Safety and Efficacy of Nivolumab in Patients With Advanced Non-small-cell Lung Cancer Treated Beyond Progression. Clin Lung Cancer. 2019 May;20(3):178-185.e2. doi: 10.1016/j.cllc.2019.02.001. Epub 2019 Feb 27. PMID 30910574
- [Background] Schadendorf D, Hodi FS, Robert C, Weber JS, Margolin K, Hamid O, Patt D, Chen TT, Berman DM, Wolchok JD. Pooled Analysis of Long-Term Survival Data From Phase II and Phase III Trials of Ipilimumab in Unresectable or Metastatic Melanoma. J Clin Oncol. 2015 Jun 10;33(17):1889-94. doi: 10.1200/JCO.2014.56.2736. Epub 2015 Feb 9. PMID 25667295
- [Background] Socinski MA, Jotte RM, Cappuzzo F, Orlandi F, Stroyakovskiy D, Nogami N, Rodriguez-Abreu D, Moro-Sibilot D, Thomas CA, Barlesi F, Finley G, Kelsch C, Lee A, Coleman S, Deng Y, Shen Y, Kowanetz M, Lopez-Chavez A, Sandler A, Reck M; IMpower150 Study Group. Atezolizumab for First-Line Treatment of Metastatic Nonsquamous NSCLC. N Engl J Med. 2018 Jun 14;378(24):2288-2301. doi: 10.1056/NEJMoa1716948. Epub 2018 Jun 4. PMID 29863955
- [Background] Stewart R, Morrow M, Hammond SA, Mulgrew K, Marcus D, Poon E, Watkins A, Mullins S, Chodorge M, Andrews J, Bannister D, Dick E, Crawford N, Parmentier J, Alimzhanov M, Babcook JS, Foltz IN, Buchanan A, Bedian V, Wilkinson RW, McCourt M. Identification and Characterization of MEDI4736, an Antagonistic Anti-PD-L1 Monoclonal Antibody. Cancer Immunol Res. 2015 Sep;3(9):1052-62. doi: 10.1158/2326-6066.CIR-14-0191. Epub 2015 May 5. PMID 25943534
- [Background] Tarhini AA, Kirkwood JM. Tremelimumab (CP-675,206): a fully human anticytotoxic T lymphocyte-associated antigen 4 monoclonal antibody for treatment of patients with advanced cancers. Expert Opin Biol Ther. 2008 Oct;8(10):1583-93. doi: 10.1517/14712598.8.10.1583. PMID 18774925
- [Background] Topalian SL, Hodi FS, Brahmer JR, Gettinger SN, Smith DC, McDermott DF, Powderly JD, Carvajal RD, Sosman JA, Atkins MB, Leming PD, Spigel DR, Antonia SJ, Horn L, Drake CG, Pardoll DM, Chen L, Sharfman WH, Anders RA, Taube JM, McMiller TL, Xu H, Korman AJ, Jure-Kunkel M, Agrawal S, McDonald D, Kollia GD, Gupta A, Wigginton JM, Sznol M. Safety, activity, and immune correlates of anti-PD-1 antibody in cancer. N Engl J Med. 2012 Jun 28;366(26):2443-54. doi: 10.1056/NEJMoa1200690. Epub 2012 Jun 2. PMID 22658127
- [Background] Topalian SL, Sznol M, McDermott DF, Kluger HM, Carvajal RD, Sharfman WH, Brahmer JR, Lawrence DP, Atkins MB, Powderly JD, Leming PD, Lipson EJ, Puzanov I, Smith DC, Taube JM, Wigginton JM, Kollia GD, Gupta A, Pardoll DM, Sosman JA, Hodi FS. Survival, durable tumor remission, and long-term safety in patients with advanced melanoma receiving nivolumab. J Clin Oncol. 2014 Apr 1;32(10):1020-30. doi: 10.1200/JCO.2013.53.0105. Epub 2014 Mar 3. PMID 24590637
- [Background] Wang DD, Zhang S, Zhao H, Men AY, Parivar K. Fixed dosing versus body size-based dosing of monoclonal antibodies in adult clinical trials. J Clin Pharmacol. 2009 Sep;49(9):1012-24. doi: 10.1177/0091270009337512. Epub 2009 Jul 20. PMID 19620385
- [Background] Wang E, Kang D, Bae KS, Marshall MA, Pavlov D, Parivar K. Population pharmacokinetic and pharmacodynamic analysis of tremelimumab in patients with metastatic melanoma. J Clin Pharmacol. 2014 Oct;54(10):1108-16. doi: 10.1002/jcph.309. Epub 2014 Apr 23. PMID 24737343
- [Background] Wolchok JD, Kluger H, Callahan MK, Postow MA, Rizvi NA, Lesokhin AM, Segal NH, Ariyan CE, Gordon RA, Reed K, Burke MM, Caldwell A, Kronenberg SA, Agunwamba BU, Zhang X, Lowy I, Inzunza HD, Feely W, Horak CE, Hong Q, Korman AJ, Wigginton JM, Gupta A, Sznol M. Nivolumab plus ipilimumab in advanced melanoma. N Engl J Med. 2013 Jul 11;369(2):122-33. doi: 10.1056/NEJMoa1302369. Epub 2013 Jun 2. PMID 23724867
- [Background] Yuan J, Adamow M, Ginsberg BA, Rasalan TS, Ritter E, Gallardo HF, Xu Y, Pogoriler E, Terzulli SL, Kuk D, Panageas KS, Ritter G, Sznol M, Halaban R, Jungbluth AA, Allison JP, Old LJ, Wolchok JD, Gnjatic S. Integrated NY-ESO-1 antibody and CD8+ T-cell responses correlate with clinical benefit in advanced melanoma patients treated with ipilimumab. Proc Natl Acad Sci U S A. 2011 Oct 4;108(40):16723-8. doi: 10.1073/pnas.1110814108. Epub 2011 Sep 20. PMID 21933959
- [Background] Zhang C, Wu S, Xue X, Li M, Qin X, Li W, Han W, Zhang Y. Anti-tumor immunotherapy by blockade of the PD-1/PD-L1 pathway with recombinant human PD-1-IgV. Cytotherapy. 2008;10(7):711-9. doi: 10.1080/14653240802320237. PMID 18841514
- [Background] Zhang S, Shi R, Li C, Parivar K, Wang DD. Fixed dosing versus body size-based dosing of therapeutic peptides and proteins in adults. J Clin Pharmacol. 2012 Jan;52(1):18-28. doi: 10.1177/0091270010388648. Epub 2011 Jan 13. PMID 21233304
- [Background] Zou W, Chen L. Inhibitory B7-family molecules in the tumour microenvironment. Nat Rev Immunol. 2008 Jun;8(6):467-77. doi: 10.1038/nri2326. PMID 18500231
- See also: Related Info — http://www.cr-technology.com/fort/